CLINICAL TRIAL: NCT01569503
Title: The Anti-inflammatory Effect of Vagus Nerve Stimulation (VNS): a New Approach in the Treatment of Crohn's Disease
Brief Title: Vagus Nerve Stimulation a New Approach in the Treatment of Crohn's Disease
Acronym: VNS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université Joseph Fourier (Other); CRSSA : Centre Recherche Service Santé Armée (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC11/12
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2017-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; VNS; vagus nerve stimulation; inflammation; Inflammatory bowel diseases; TNF
MeSH Terms: conditions — Crohn Disease; Inflammation; Inflammatory Bowel Diseases | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VSN (Experimental): VNS therapy
  Interventions: Device: vagus nerve stimulation (VNS)

INTERVENTIONS:
Device: vagus nerve stimulation (VNS) — VNS therapy consists of an implanted pacemaker-like device that delivers mild, intermittently pulsed signals to the patient's left vagus nerve. Roughly the size of a small pocket-watch and weighing less than one ounce, the pulse generator is implanted in the patient's left chest area. A thin thread-like wire, attached to the generator, runs under the skin to the left vagus nerve in the neck

SUMMARY:
The purpose of this study is to determine whether (VNS) Vagus Nerve Stimulation , is effective in the treatment of Crohn's disease.

DETAILED DESCRIPTION:
Inflammatory bowel diseases or IBD (Crohn's disease and ulcerative colitis) are chronic inflammatory diseases involving the digestive tract, in particular the small bowel and/or the recto-colon. IBD represent a public health problem in Gastroenterology. The etiopathogeny of IBD is multifactorial involving immunological, genetic, infectious and environmental factors. An overarching hypothesis is that an unbalance of the autonomic nervous system, represented by the sympathetic and parasympathetic nervous system (e.g. the vagus nerve) is part of the mechanisms underlying the pathophysiology of IBD. A dysautonomia has been observed in IBD patients and we have recently demonstrated that this dysautonomia was linked to psychological coping, in particular in Crohn's disease. Classically, the vagus nerve, a mixed nerve, has an anti-inflammatory role through its central afferents which secondarily stimulate the hypothalamic-pituitary adrenal axis. Recent data have shown that the anti-inflammatory properties of the vagus nerve also involve peripheral efferents via an interaction of acetylcholine with nicotinic receptors leading to an inhibition of TNF release by macrophages. Vagus nerve stimulation (VNS) is currently used for the treatment of some forms of epilepsy in Human via a stimulation of vagal afferents. We have recently validated a model of chronic VNS (3h/d for 5 days) in freely moving rats by stimulating vagal efferents and we have studied the anti-inflammatory properties of VNS in an experimental model of colitis in rats. VNS significantly decreased body weight loss due to colitis and had an anti-inflammatory effect by decreasing a multivariate index of inflammation. To date, medical treatment of IBD (e.g. 5-aminosalicylates, corticosteroids, immunosuppressives or biotherapies i.e. anti-TNF) is only suspensive. The aim of our project is to propose another type of anti-inflammatory treatment based on neurostimulation of vagal efferents. For this purpose, we aim to perform a pilot study in 10 patients with moderate to severe Crohn's disease despite a reference treatment (corticosteroids and/or immunosuppressives) using the anti-inflammatory properties of VNS as an alternative to anti-TNF therapy. Central and peripheral effect of VNS will be also evaluated by electroencephalographic and sympatho-vagal (heart rate variability) recordings. The finality, at term, is to use VNS as an alternative to the conventional anti-TNF therapy not devoid of side effects, in particular infectious, with the advantage to use an intrinsic anti-inflammatory (anti-TNF) system and to take cover of problems of adherence to treatment which are frequently observed in the medical treatment of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD involving the ileo-colon, diagnosed for at least 3 months prior to screening in flare (220<CDAI<450) of their disease despite a treatment reference (corticosteroids and/or immunosuppressives) with a stable dose will be included
* CRP>5mg/l and/or fecal calprotectin <100µg/l
* CDEIS > 7 (Crohn's disease endoscopic index of severity)
* Consenting patient

Exclusion Criteria:

* Known cardiac pathology
* VNS contraindication
* Anoperineal CD only or associated with ileocolic lesion
* Diagnosis of indeterminate colitis, positive stool culture for enteric pathogens
* CD Surgery within 3 months before screening
* Short small intestine (<1m)
* Koenig syndrome
* Intra-abdominal abscess
* Fistula with clinical or radiological abscess evidence
* Anoperineal CD with or without rectal involvement
* Ileostomy, colostomy, enteral or parenteral feeding
* Clinical condition medically or surgically unstable that, at the discretion of the investigator would not be compatible with the patient's participation in the study
* Any recent neoplasia, in the year prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical remission 12 months after initiation of VNS | 12 months after initiation of VNS
  Clinical remission at 12 months :
  1. Patient without corticoids or a dose of 20mg without dose adjustment (stable treatment) and without anti-TNF,
  2. CDAI <150 or CDAI has dropped by at least 70 or 100 points (Δ70, Δ100) compared with the baseline CDAI
  3. Stable immunosuppressive therapy.

SECONDARY OUTCOMES:
Clinical remission 6 months after initiation of VNS | 6 months after initiation of VNS
  Clinical remission at 6 months :
  1. Patient without corticoids or a dose of 20mg without dose adjustment (stable treatment) and without anti-TNF,
  2. CDAI <150 or CDAI has dropped by at least 70 or 100 points (Δ70, Δ100) compared with the baseline CDAI
  3. Stable immunosuppressive therapy
VNS tolerance | 12 months
  Description and frequency of adverse events
Assessment of VNS effectiveness with biological markers | 12 months
  Assessment of VNS effectiveness with biological markers of the pro-and anti-inflammatory status
Endoscopic and ultrasound Assessment of VNS effectiveness | 12 months
  Endoscopy : CDEIS (Crohn's Disease Endoscopic Index of Severity) Ultrasound : score Migaleddu V. and al, 2009
Assessment of the central effects of VNS | At 6 weeks, at 6 months, at 12 months
  Evolution of :
  * Sleep cycle : duration of sleep stages, sleep latency, latency between the different sleep stages.
  * High-resolution Electroencephalogram (EEG): Spatiotemporal evolution of the spectral density of EEG power in the different frequency bands
  * Correlation between high-resolution EEG markers of autonomic nervous system
Evaluation of peripheral effects of VNS on sympatho-vagal balance | 6 weeks, 6 months, 12 months
  Evolution of cardiac variability markers using time and frequency analysis of electrocardiogram :
  * Frequency Analysis : LH, HF, LF/HF
  * Time analysis : RMS-SD, pNN50, NN50, average cardiac rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BONAZ, MD, PHD, Principal Investigator — Grenoble university hsopital
Locations (1):
- Grenoble university hospital, Grenoble, Isere, France

REFERENCES:
- [Background] Meregnani J, Clarencon D, Vivier M, Peinnequin A, Mouret C, Sinniger V, Picq C, Job A, Canini F, Jacquier-Sarlin M, Bonaz B. Anti-inflammatory effect of vagus nerve stimulation in a rat model of inflammatory bowel disease. Auton Neurosci. 2011 Feb 24;160(1-2):82-9. doi: 10.1016/j.autneu.2010.10.007. Epub 2010 Nov 11. PMID 21071287
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541